CLINICAL TRIAL: NCT03809052
Title: GB1211 - A Randomised, Double-Blind, Placebo-Controlled, First-In-Human, Study of Orally Administered GB1211 to Evaluate the Safety, Tolerability, and PK of Single Ascending Doses (SAD) and Multiple Ascending Doses (MAD) in Healthy Subjects
Brief Title: A First in Human Study to Evaluate the Safety, Tolerability and PK of GB1211 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galecto Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: GB1211-001; 2018-003914-41 (EudraCT Number); Covance Study Number: 8392356 (Other: Covance)
Record Dates: First submitted 2018-12-07; First posted 2019-01-18 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2019-01

CONDITIONS: Safety and Tolerability
Keywords: GB1211; Phase 1; First Time in Human; Safety; Tolerability; Pharmacokinetics; Single Ascending Dose (SAD); Multiple Ascending Dose (MAD); Healthy Volunteers; Nonalcoholic Steatohepatitis (NASH); Liver Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Part A: 56 subjects will be studied in 7 cohorts (Cohorts A1 to A7) Part B: 22 subjects will be studied in 2 cohorts (Cohorts B1 to B2)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- A1 - 5 mg GB1211 single dose and Placebo (Experimental): 6 healthy subjects are administered 5 mg of GB1211 capsules orally as a single dose in the fasted state. 2 subjects receive placebo. 2 subjects (1 active and 1 placebo) will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  Interventions: Drug: GB1211
- A2 - 20 mg GB1211 single dose and Placebo (Experimental): 6 healthy subjects are administered 20 mg of GB1211 capsules orally as a single dose in the fasted state. 2 subjects receive placebo. 2 subjects (1 active and 1 placebo) will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  Interventions: Drug: GB1211
- A3 - 50 mg GB1211 single dose (food effect cohort) and Placebo (Experimental): 6 healthy subjects are administered 50 mg of GB1211 capsules orally as a single dose. 2 subjects receive placebo. 2 subjects (1 active and 1 placebo) will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion. Each subject will participate in 2 treatment periods separated by a minimum of 7 days. In Treatment Period 1 doses will be administered in the fasted state, in Treatment Period 2 doses will be administered 30 minutes after the start of a high fat breakfast. Subjects will receive the same treatment in both periods.
  Interventions: Drug: GB1211
- A4 - 100 mg GB1211 single dose and Placebo (Experimental): 6 healthy subjects are administered 100 mg of GB1211 capsules orally as a single dose in the fasted state. 2 subjects receive placebo. 2 subjects (1 active and 1 placebo) will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  Interventions: Drug: GB1211
- A5 - 200 mg GB1211 single dose and Placebo (Experimental): 6 healthy subjects are administered 200 mg of GB1211 capsules orally as a single dose in the fasted state. 2 subjects receive placebo. 2 subjects (1 active and 1 placebo) will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  Interventions: Drug: GB1211
- B1 - GB1211 multiple ascending doses, 50mg BID and Placebo (Experimental): GB1211 administered orally twice daily over 10 days. 8 healthy subjects received GB1211 and 3 subjects will receive placebo. Following review of data in Part A (Cohorts A1 to A6), subjects received twice daily (BID) doses under fasted conditions on Days 1 to 9, inclusive, and a final single dose administration on the morning of Day 10 in accordance with the randomisation schedule.
  Interventions: Drug: GB1211
- B2 - GB1211 multiple ascending doses, 100mg BID and Placebo (Experimental): GB1211 administered orally twice daily over 10 days. 8 healthy subjects received GB1211 and 3 subjects will receive placebo. Following review of data in Part A (Cohorts A1 to A6), subjects received twice daily (BID) doses under fasted conditions on Days 1 to 9, inclusive, and a final single dose administration on the morning of Day 10 in accordance with the randomisation schedule..
  Interventions: Drug: GB1211
- A6 - 50mg GB1211 single dose and Placebo (Experimental): 8 healthy subjects are administered 50 mg (10 x 5mg capsules) or placebo without sentinel dosing. Optional cohort, as was added following dose-escalation analysis.
  Interventions: Drug: GB1211
- A7 - 400 mg GB1211 single dose and Placebo (Experimental): 8 healthy subjects are administered 400 mg (8 x 50mg capsules) or placebo without sentinel dosing. Optional cohort, as was added following dose-escalation analysis.
  Interventions: Drug: GB1211
- Part A - Placebo for GB1211 (Experimental): In Part A - 2 subjects from each arm (A1-A5) will receive placebo.
  Interventions: Drug: Placebo
- Part B - Placebo for GB1211 (BID) (Experimental): Part B - 3 subjects from each arm B1 and B2 will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GB1211 — Hard capsules for oral use
  Arms: A1 - 5 mg GB1211 single dose and Placebo; A2 - 20 mg GB1211 single dose and Placebo; A3 - 50 mg GB1211 single dose (food effect cohort) and Placebo; A4 - 100 mg GB1211 single dose and Placebo; A5 - 200 mg GB1211 single dose and Placebo; A6 - 50mg GB1211 single dose and Placebo; A7 - 400 mg GB1211 single dose and Placebo; B1 - GB1211 multiple ascending doses, 50mg BID and Placebo; B2 - GB1211 multiple ascending doses, 100mg BID and Placebo
Drug: Placebo — Hard capsules for oral use
  Other Names: GB1211
  Arms: Part A - Placebo for GB1211; Part B - Placebo for GB1211 (BID)

SUMMARY:
This was a Phase 1, randomized, double-blind, placebo-controlled, first-in-human study in which the safety, tolerability, and pharmacokinetics of orally administered GB1211 will be evaluated in healthy adult subjects and adult subjects with indication of suspected Nonalcoholic steatohepatitis (NASH) and liver fibrosis.

DETAILED DESCRIPTION:
The study consisted of 2 parts: a SAD phase (Part A) which enrolled a total of 5 cohorts of healthy subjects and a MAD phase (Part B) which enrolled 2 cohorts of healthy subjects. Two additional cohorts A6 and A7, were added following dose escalation analysis.

The planned optional Part C was to include a multiple-dose cohort of 25 subjects with suspected NASH and liver fibrosis (Cohort C1). However, Part C of the study was not performed as per Sponsor's decision.

ELIGIBILITY:
Inclusion Criteria:

Subjects for Parts A and B must satisfy all of the following criteria at the Screening visit unless otherwise stated:

1. Males or females, of any race, between 18 and 55 years of age (60 years for Part B), inclusive.
2. Body mass index (BMI) of 18.0 to 32.0 kg/m^2 (inclusive) with a minimum body weight of 50 kg.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations
4. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception as detailed further in the protocol.
5. Male subjects must agree to refrain from sperm donation and females should refrain from ova donation from the date of Check-in (Day -1) until 90 days after the Follow-up visit.
6. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Subjects for Parts C must satisfy all of the following criteria at the Screening visit unless otherwise stated:

1. Males or females, of any race, between 18 and 60 years of age, inclusive.
2. Body mass index (BMI) of ≥ 25.0 and ≤ 38.0 kg/m^2.
3. Documented history of fatty liver within the last 24 weeks by one of the following: magnetic resonance imaging (MRI) suggesting liver fat ≥ 8%, ultrasound (US) indicating fatty liver, or Fibroscan Controlled Attenuation Parameter (CAP) > 270 dB/m. In subjects without a documented history of fatty liver, a Fibroscan CAP or US can be performed at Screening. Subjects with Fibroscan CAP > 270 dB/m or US indicating fatty liver are eligible.
4. Metabolic syndrome (Adult Treatment Panel III definition) or T2DM (defined as stable diabetes with glycosylated haemoglobin [HbA1c] ≤ 9.5%).
5. Alanine aminotransferase (ALT) ≥ 20 U/L for females and ≥ 30 U/L for males at Screening.
6. Fibroscan ≥ 7 KPa and < 13 KPa, or Fibrosis-4 (FIB-4) index ≥ 1.1 and <3.25.
7. Females of nonchildbearing potential defined as permanently sterile (ie, due to hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy) or postmenopausal (defined as at least 12 months postcessation of menses without an alternative medical cause and follicle-stimulating hormone [FSH] level ≥ 40 mIU/mL). Males will agree to use contraception as detailed in protocol.
8. Male subjects must agree to refrain from sperm donation and females should refrain from ova donation from the date of Check-in (Day -1) until 90 days after the Follow-up visit.
9. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

Subjects from Part A & B will be excluded from the study if they satisfy any of the following criteria at the Screening visit unless otherwise stated:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.

3 (Part A). Any of the following: a. QTcF > 450 msec confirmed by repeat measurement. b. QRS duration > 110 msec confirmed by repeat measurement. c. PR interval > 220 msec confirmed by repeat measurement. d. findings which would make QTc measurements difficult or QTc data uninterpretable. e. history of additional risk factors for torsades de pointes (eg, heart failure, hypokalaemia, family history of long QT syndrome).

3 (Part B). Clinically significant ECG abnormalities or QTcF greater than 450 msec for males and 470 msec for females at either Screening or Day 1 predose, or any prior history of QT abnormality.

4. History of alcoholism or drug/chemical abuse within 1 year prior to Check-in.

5. Positive hepatitis panel and/or positive human immunodeficiency virus (HIV) test.

6. Participation in a clinical study involving administration of an investigational agent or vaccine (new chemical entity) or having received a biological product in the past 90 days prior to dosing.

7. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing, unless deemed acceptable by the Investigator (or designee).

8. Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee).

9. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in, or positive cotinine at Screening or Check-in.

10. Receipt of blood products within 2 months prior to Check-in and donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.

11. Subject who, in the opinion of the Investigator (or designee), should not participate in this study.

Subjects from Part C will be excluded from the study if they satisfy any of the following criteria at the Screening visit unless otherwise stated:

1. If diabetic and diabetes is other than T2DM.
2. Subjects, who have had bariatric surgery of any kind or, in the opinion of the Investigator, have experienced a clinically significant change in body weight within the 3 months prior to Screening.
3. History of any known serious disease (such as cancer, except skin basocellular carcinomas, major infection, clinically significant gastrointestinal disorder, major autoimmune disease) or other disease which in the Investigator's opinion would exclude the patient from the study.
4. The following clinical laboratory results at Screening: -Total Bilirubin > 2 × ULN, ALT > 155 U/L for females and > 185 U/L for males, AST > 155 U/L for females and > 200 U/L for males
5. Other abnormal clinical laboratory values that are considered clinically significant for this population.
6. Clinically significant ECG abnormalities or QTcF greater than 450 msec for males and 470 msec for females at either Screening or Day 1 predose, or any prior history of QT abnormality.
7. History of alcoholism or drug/chemical abuse within 1 year prior to Check-in.
8. Alcohol consumption of > 14 units per week for males and for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
9. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at Screening or Check-in.
10. Positive hepatitis panel and/or positive HIV test .
11. A creatinine clearance of less than 50 mL/min (as calculated by Cockcroft-Gault equation) or estimated glomerular filtration rate (eGFR) < 60 mL/[min*1.73 m²] at Screening.
12. Subject taking any antidiabetic medications, with the exception of metformin, sulfonylureas, gliptins, and sodium/glucose co-transporter 2 inhibitors, within 3 months prior to Screening.
13. Use of any of the following non-permitted medication within 6 months prior to Screening: amiodarone, bile salt chelators, methotrexate, pharmacological doses of systemic corticosteroids for at least 2 consecutive weeks, or any other medications known to affect liver function.
14. Have previously completed or withdrawn from this study investigating GB1211, and have previously received the investigational product.
15. Subject who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ashley Brooks, MBChB, Principal Investigator — Covance; Dr Bertil Lindmark MD PHD, Chief Medical Officer, Study Chair — Galecto Biotech AB
Locations (1):
- (For Parts A and B) Covance Clinical Research Unit Ltd, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aslanis V, Slack RJ, MacKinnon AC, McClinton C, Tantawi S, Gravelle L, Nilsson UJ, Leffler H, Brooks A, Khindri SK, Marshall RP, Pedersen A, Schambye H, Zetterberg F. Safety and pharmacokinetics of GB1211, an oral galectin-3 inhibitor: a single- and multiple-dose first-in-human study in healthy participants. Cancer Chemother Pharmacol. 2023 Mar;91(3):267-280. doi: 10.1007/s00280-023-04513-y. Epub 2023 Mar 13. PMID 36914828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 78 subjects entered the study and were randomised to treatment, with 56 subjects in Part A and 22 subjects in Part B.
Groups:
- A1 - 5 mg GB1211 Single Dose: 6 healthy subjects are administered 5 mg of GB1211 capsules orally as a single dose in the fasted state. 1 subject will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  GB1211: Hard capsules for oral use
- A2 - 20 mg GB1211 Single Dose: 6 healthy subjects are administered 20 mg of GB1211 capsules orally as a single dose in the fasted state. 1 subject will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  GB1211: Hard capsules for oral use
- A3 - 50 mg GB1211 Single Dose (Food Effect Cohort): 6 healthy subjects are administered 50 mg of GB1211 capsules orally as a single dose in the fasted state. 1 subject will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  Each subject will participate in 2 treatment periods separated by a minimum of 7 days. In Treatment Period 1 doses will be administered in the fasted state, in Treatment Period 2 doses will be administered 30 minutes after the start of a high fat breakfast. Subjects will receive the same treatment in both periods.
  GB1211: Hard capsules for oral use
- A4 - 100 mg GB1211 Single Dose: 6 healthy subjects are administered 100 mg of GB1211 capsules orally as a single dose in the fasted state. 1 subject will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  GB1211: Hard capsules for oral use
- A5 - 200 mg GB1211 Single Dose: 6 healthy subjects are administered 200 mg of GB1211 capsules orally as a single dose in the fasted state. 1 subject will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  GB1211: Hard capsules for oral use
- A6 - 50mg GB1211 Single Dose: 6 healthy subjects are administered 50 mg without sentinel dosing. Optional cohort, as was added following dose-escalation analysis.
  GB1211: Hard capsules for oral use
- A7 - 400 mg GB1211 Single Dose: 6 healthy subjects are administered 400 mg without sentinel dosing. Optional cohort, as was added following dose-escalation analysis.
  GB1211: Hard capsules for oral use
- Part A - Placebo GB1211: In Part A, 14 subjects will receive placebo in total.
  Placebo: Hard capsules for oral use
- B1 - GB1211 Multiple Ascending Doses, 50mg BID: GB1211 50 mg administered orally twice daily over 10 days. 8 healthy subjects received GB1211. Following review of data in Part A (Cohorts A1 to A6), subjects received twice daily (BID) doses under fasted conditions on Days 1 to 9, inclusive, and a final single dose administration on the morning of Day 10 in accordance with the randomisation schedule.
  GB1211: Hard capsules for oral use
- B2 - GB1211 Multiple Ascending Doses, 100mg BID: GB1211 100 mg administered orally twice daily over 10 days. 8 healthy subjects received GB1211. Following review of data in Part A (Cohorts A1 to A6), subjects received twice daily (BID) doses under fasted conditions on Days 1 to 9, inclusive, and a final single dose administration on the morning of Day 10 in accordance with the randomisation schedule.
  GB1211: Hard capsules for oral use
- Part B - PLacebo GB1211 (BID): In Part B, 6 subjects will receive placebo in total.
  Placebo: Hard capsules for oral use
Period: Overall Study
Arm/Group | A1 - 5 mg GB1211 Single Dose | A2 - 20 mg GB1211 Single Dose | A3 - 50 mg GB1211 Single Dose (Food Effect Cohort) | A4 - 100 mg GB1211 Single Dose | A5 - 200 mg GB1211 Single Dose | A6 - 50mg GB1211 Single Dose | A7 - 400 mg GB1211 Single Dose | Part A - Placebo GB1211 | B1 - GB1211 Multiple Ascending Doses, 50mg BID | B2 - GB1211 Multiple Ascending Doses, 100mg BID | Part B - PLacebo GB1211 (BID)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 8 | 8 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 8 | 8 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- A3 - 50 mg GB1211 Single Dose (Food Effect Cohort): 6 healthy subjects are administered 50 mg of GB1211 capsules orally as a single dose in the fasted state. 1 subject will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  GB1211: Hard capsules for oral use
- Part A - Placebo for GB1211: In Part A, 14 subjects will receive placebo in total.
  Placebo: Hard capsules for oral use Placebo: Hard capsules for oral use
- B1 - GB1211 Multiple Ascending Doses, 50mg BID: GB1211 50mg administered orally twice daily over 10 days. 8 healthy subjects received GB1211. Following review of data in Part A (Cohorts A1 to A6), subjects received twice daily (BID) doses under fasted conditions on Days 1 to 9, inclusive, and a final single dose administration on the morning of Day 10 in accordance with the randomisation schedule.
  GB1211: Hard capsules for oral use
- B2 - GB1211 Multiple Ascending Doses, 100mg BID: GB1211 100mg administered orally twice daily over 10 days. 8 healthy subjects received GB1211. Following review of data in Part A (Cohorts A1 to A6), subjects received twice daily (BID) doses under fasted conditions on Days 1 to 9, inclusive, and a final single dose administration on the morning of Day 10 in accordance with the randomisation schedule.
  GB1211: Hard capsules for oral use
- Part B - Placebo for GB1211 (BID): In Part B, 6 subjects will receive placebo in total.
  Placebo: Hard capsules for oral use
  Placebo: Hard capsules for oral use
- Total: Total of all reporting groups
Arm/Group | A1 - 5 mg GB1211 Single Dose | A2 - 20 mg GB1211 Single Dose | A3 - 50 mg GB1211 Single Dose (Food Effect Cohort) | A4 - 100 mg GB1211 Single Dose | A5 - 200 mg GB1211 Single Dose | A6 - 50mg GB1211 Single Dose | A7 - 400 mg GB1211 Single Dose | Part A - Placebo for GB1211 | B1 - GB1211 Multiple Ascending Doses, 50mg BID | B2 - GB1211 Multiple Ascending Doses, 100mg BID | Part B - Placebo for GB1211 (BID) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 8 | 8 | 6 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (7.4) | 38 (12.8) | 28 (8.0) | 35 (9.2) | 36 (12.8) | 34 (13.5) | 39 (11.3) | 37 (13.3) | 42 (12.6) | 37 (11.6) | 39 (8.1) | 36 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 1 | 1 | 2 | 2 | 6 | 3 | 3 | 2 | 27
  Male | 3 | 4 | 4 | 5 | 5 | 4 | 4 | 8 | 5 | 5 | 4 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 8 | 8 | 6 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 5
  White | 4 | 4 | 5 | 5 | 6 | 5 | 6 | 11 | 8 | 8 | 6 | 68
  More than one race | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilogram] | 75.9 (7.27) | 77.9 (19.03) | 71.4 (7.87) | 75.1 (13.94) | 73.7 (11.61) | 73.3 (16.72) | 79.7 (12.63) | 81.3 (12.82) | 85.4 (17.20) | 76.8 (9.52) | 70.9 (13.24) | 76.5 (12.9)
Height [Mean (Standard Deviation); unit: centimeter] | 172.3 (10.31) | 171.7 (9.65) | 169.8 (5.00) | 175.3 (5.20) | 174.7 (8.45) | 176.2 (12.86) | 173.7 (8.12) | 173.6 (10.26) | 178.9 (7.62) | 173.4 (4.21) | 175.2 (5.71) | 174.1 (7.9)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (4.48) | 26.1 (3.91) | 24.8 (2.73) | 24.5 (4.63) | 24.1 (3.25) | 23.3 (2.86) | 26.2 (1.90) | 26.9 (3.06) | 26.5 (3.78) | 25.5 (2.35) | 23.0 (3.50) | 25.2 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With of Adverse Events (AEs)
Description: The number of participants in each arm that report Adverse Events (AEs)
Time Frame: Up to 5-7 days post final dose (Part A: Single dose), Part B: 6-7 weeks
Population: All subjects in part A and B were included in the safety populations. The safety population will include all subjects who received at least 1 dose of study treatment (GB1211 or placebo). Safety parameters will be listed and summarised using descriptive statistics. No formal statistical analysis of safety data is planned.
Measure: Number; unit: Count of Participants
Groups:
- A3 - 50 mg GB1211 Single Dose (Food Effect Cohort): 6 healthy subjects are administered 50 mg of GB1211 capsules orally as a single dose. 2 subjects receive placebo. 2 subjects (1 active and 1 placebo) will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion. Each subject will participate in 2 treatment periods separated by a minimum of 7 days. In Treatment Period 1 doses will be administered in the fasted state, in Treatment Period 2 doses will be administered 30 minutes after the start of a high fat breakfast. Subjects will receive the same treatment in both periods.
  GB1211: Hard capsules for oral use
- Part A - Placebo for GB1211: In Part A, 14 subjects will receive placebo in total.
  Placebo: Hard capsules for oral use
- Part B - Placebo for GB1211 (BID): In Part B, 6 subjects will receive placebo in total.
  Placebo: Hard capsules for oral use
Arm/Group | A1 - 5 mg GB1211 Single Dose | A2 - 20 mg GB1211 Single Dose | A3 - 50 mg GB1211 Single Dose (Food Effect Cohort) | A4 - 100 mg GB1211 Single Dose | A5 - 200 mg GB1211 Single Dose | A6 - 50mg GB1211 Single Dose | A7 - 400 mg GB1211 Single Dose | Part A - Placebo for GB1211 | B1 - GB1211 Multiple Ascending Doses, 50mg BID | B2 - GB1211 Multiple Ascending Doses, 100mg BID | Part B - Placebo for GB1211 (BID)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 8 | 8 | 6
Count of Participants | 3 | 1 | 1 | 1 | 0 | 2 | 1 | 5 | 1 | 4 | 3

ADVERSE EVENTS:
Time Frame: Up to 5-7 days post final dose (Part A: Single dose), Part B: 6-7 weeks
Groups:
- Part A - Placebo GB1211 (Fed): In Part A, 2 subjects will receive placebo in total in a fed state.
  Placebo: Hard capsules for oral use
- A3 - 50 mg GB1211 Single Dose (Period 1: Fasted)" and "A3- 50 mg GB1211 Single Dose (Period 2: Fed): 6 healthy subjects are administered 50 mg of GB1211 capsules orally as a single dose in the fasted state. 1 subject will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  GB1211: Hard capsules for oral use
- A3- 50 mg GB1211 Single Dose (Fed): 6 healthy subjects are administered 50 mg without sentinel dosing. Optional cohort, as was added following dose-escalation analysis.
  GB1211: Hard capsules for oral use
- A7 - 400 mg GB1211 Single Dose: 6 healthy subjects are administered 400 mg of GB1211 capsules orally as a single dose in the fasted state. 1 subject will be dosed at least 24 hours before the remaining subjects, where continuation to dose the remaining subjects will be at the Investigator's discretion.
  GB1211: Hard capsules for oral use
Arm/Group | Part A - Placebo for GB1211 | Part A - Placebo GB1211 (Fed) | A1 - 5 mg GB1211 Single Dose | A2 - 20 mg GB1211 Single Dose | A3 - 50 mg GB1211 Single Dose (Period 1: Fasted)" and "A3- 50 mg GB1211 Single Dose (Period 2: Fed) | A6 - 50mg GB1211 Single Dose | A3- 50 mg GB1211 Single Dose (Fed) | A4 - 100 mg GB1211 Single Dose | A5 - 200 mg GB1211 Single Dose | A7 - 400 mg GB1211 Single Dose | Part B - Placebo for GB1211 (BID) | B1 - GB1211 Multiple Ascending Doses, 50mg BID | B2 - GB1211 Multiple Ascending Doses, 100mg BID
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/14 | 1/2 | 3/6 | 1/6 | 1/6 | 1/6 | 1/6 | 1/6 | 0/6 | 1/6 | 1/6 | 4/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Placebo for GB1211 (N=14) | Part A - Placebo GB1211 (Fed) (N=2) | A1 - 5 mg GB1211 Single Dose (N=6) | A2 - 20 mg GB1211 Single Dose (N=6) | A3 - 50 mg GB1211 Single Dose (Period 1: Fasted)" and "A3- 50 mg GB1211 Single Dose (Period 2: Fed) (N=6) | A6 - 50mg GB1211 Single Dose (N=6) | A3- 50 mg GB1211 Single Dose (Fed) (N=6) | A4 - 100 mg GB1211 Single Dose (N=6) | A5 - 200 mg GB1211 Single Dose (N=6) | A7 - 400 mg GB1211 Single Dose (N=6) | Part B - Placebo for GB1211 (BID) (N=6) | B1 - GB1211 Multiple Ascending Doses, 50mg BID (N=8) | B2 - GB1211 Multiple Ascending Doses, 100mg BID (N=8)
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 — TEAEs reported at Part B Placebo group (1AE) and Part B B1 100mg BID group (2AEs) were determined to be drug related
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — The TEAE was determined to be drug-related
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — The TEAE was determined to be drug-related
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — The TEAE was determined to be drug related
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — The TEAE was determined to be drug related
Medical device site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — The TEAE was determined to be drug-related
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 — The TEAE reported at Part A Placebo group was determined to be drug related. The TEAE reported on 3 subjects from Part B B1 50mg BID group were determined to be drug related
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — The TEAE was determined to be drug-related
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — The TEAE was determined to be drug related
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — The TEAE was determined to be drug related
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 — The TEAE reported to 2 subjects was determined to be tdrug related
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — the TEAE was determined to be drug related
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — the TEAE was determined to be drug related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT03809052/SAP_000.pdf
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT03809052/Prot_001.pdf